CLINICAL TRIAL: NCT01693198
Title: Cyanobacteria Allergy in Lake Kineret
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Yigal Allon Kinneret Limnological Laboratory (Unknown)
Responsible Party: Principal Investigator, Ronit Confino-Cohen, MD, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0172-12-MMC
Record Dates: First submitted 2012-09-19; First posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Nasal Stuffiness; Sneezing; Itching
Keywords: allergy; cyanobacteria; sweet water swimming
MeSH Terms: conditions — Nasal Obstruction; Sneezing; Pruritus; Hypersensitivity | interventions — Skin Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Skin test with sterile extracts of different cyanobacteria — Skin test with sterile extracts of different cyanobacteria is performed on the volar aspect of the forearm. Typically, the results are read 15 minutes after performing the test. Test is regarded as positive when wheal of more than 3mm and flare appear within this time frame. Positive test indicates the existence of specific IgE to the extract in on skin mast cells .

SUMMARY:
People swimming or surfing in lake Kineret , sometimes complain of nasal stuffiness , sneezing and itching .Typically, it happens during or immediately after contact with the lake's water . The symptoms are compatible with immediate allergic reaction. Previous reports suggested a connection between similar symptoms and contact with different cyanobacteria (living in fresh water lakes). In this study we intend to prove the mechanism of these reactions. To prove the exact allergen that causes allergic rhinitis allergists perform skin tests with different suspected allergens. Likewise, we would like to perform skin tests to different proteins extracted from cyanobacteria collected in lake Kineret.

ELIGIBILITY:
Inclusion Criteria:

* age above 18
* exposed to Lake Keneret water by swiming or sirfing

Exclusion Criteria:

* age under 18
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of skin test to cyanobacteria | Immediately after performing the test (15 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center, Kfar Saba, Israel

REFERENCES:
- [Background] 1. Carmichael W. A world overview-One-hundred-twentyseven years of research on toxic cyanobacteria-Where do we go from here? Adv Exp Med Biol 2008;619:105-125 2. Petrus M, Culerrier R, Campistron M, Barre A, Rouge P. First case report of anaphylaxis to spirulin: identification of phycocyanin as responsible allergen. AL L ERGY (AllergyNet) 2010; 65 : 924-932N 3. Torokne A, Palovics A, and Bankine M. Allergenic (sensitization, skin and eye Irritation).Effects of freshwater Cyanobacteria-experimental evidence. Environ Toxicol 2001; 16: 512-516 4.Alster, A., Kaplan-Levy, R., Sukenik, A. & Zohary, T. Morphology and phylogeny of a non-toxic invasive Cylindrospermopsis raciborskii from a Mediterranean Lake. Hydrobiologia 2010; 639, 115-128. 5.Banker, R., Carmeli, S., Hadas, O., Teltsch, B., Porat, R. & Sukenik, A. Identification of cylindrospermopsin in Aphanizomenon ovalisporum (Cyanophyceae) isolated from Lake Kinneret, Israel. Journal of Phycology 1997; 33, 613-616. 6.Hadas, O., Pinkas, R., Malinsky-Rushansky, N., Nishri, A., Kaplan, A., Rimmer, A. & Sukenik, A. Appearance and establishment of diazotrophic cyanobacteria in Lake Kinneret, Israel. Freshwater Biology 2012; 57, 1214-1227. 7. Bernstein JA, Ghosh D, Levin LS, Zheng S, Carmichael W, Lummus Z, Bernstein IL. Cyanobacteria: an unrecognized ubiquitous sensitizing allergen? Allergy Asthma Proc. 2011;32:106-110 8.Törökné, A., Asztalos, M., Bánkiné, M., Bickel, H., Borbély, G., Carmeli, S., Codd, G.A., Fastner, J., Huang, Q., Humpage, A., Metcalf, J.S., Rábai, E., Sukenik, A., Surányi, G., Vasas, G. & Weiszfeiler, V. Interlaboratory comparison trial on cylindrospermopsin measurement. Analytical Biochemistry 2004; 332, 280-284. 9.Lawton, L.A., Edwards, C. & Codd, G.A. Extraction and high-performance liquid chromatographic method for the determination of microcystins in raw and treated waters. Analyst 1994; 119, 1525-1530